CLINICAL TRIAL: NCT01899235
Title: The Treatment of Coronary De-novo Lesions With the Elutax Paclitaxel-eluting Balloon Alone, a Pilot Study
Acronym: EXPEL
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Slow recruitment
Sponsor: Aalborg University Hospital (Other)
Collaborators: Aachen Resonance GmbH (Industry)
Responsible Party: Principal Investigator, Svend Eggert Jensen, Associate professor, MD, PhD, Aalborg University Hospital
Purpose: Treatment
Other Study IDs: N-20110015
Record Dates: First submitted 2013-07-11; First posted 2013-07-15 (Estimated); Last update posted 2014-03-18 (Estimated); Status verified 2014-03

CONDITIONS: Stable Angina; Coronary Stenosis
MeSH Terms: conditions — Angina, Stable; Coronary Stenosis | interventions — Drug-Eluting Stents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stent (Active Comparator): drug eluting stent (Resolute)
  Interventions: Device: drug eluting stent
- drug eluting balloon (Experimental): drug eluting balloon (Elutax)
  Interventions: Device: drug eluting balloon

INTERVENTIONS:
Device: drug eluting balloon
  Arms: drug eluting balloon
Device: drug eluting stent
  Arms: Stent

SUMMARY:
A randomised open-label pilot study to assess the safety and efficacy of treatment with a drug eluting balloon alone in coronary de novo lesions). Elective patients requiring PCI to coronary de novo lesions in vessels 2.5 mm - 4.0 mm.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18years old
* Stable angina symptoms
* Elective treatment to coronary lesion
* Reference vessel diameters of ≥ 2.5mm and ≤ 4.0 mm on visual inspection

Exclusion Criteria:

* Left main stem lesion
* Bifurcation lesions
* Acute coronary syndrome (UAP, NSTEMI, STEMI)
* Cardiogenic shock
* Chronic total occlusion
* Additional lesions requiring PCI
* Platelet count ≤ 50 x 109/mm3
* Left ventricular ejection fraction ≤ 30%
* Patient life expectancy less than 12 months
* Known allergies to aspirin, clopidogrel, prasugrel, heparin, stainless steel, intravenous contrast (severe), or paclitaxel
* Participation in another investigational drug or device study
* Patient unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2011-05; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Major adverse cardiac events | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Aalborg University Hospital, Aalborg, Denmark